CLINICAL TRIAL: NCT07266311
Title: Clinical Study on the Safety and Efficacy of CAR T-cell Therapy for Claudin18.2 Positive Advanced Solid Malignant Tumors
Brief Title: CAR-T for Claudin18.2 Positive Solid Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chengdu Ucello Biotechnology Co., Ltd. (Industry)
Collaborators: The General Hospital of Western Theater Command (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T_CLDN18.2
Record Dates: First submitted 2025-11-22; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Claudin18.2 Positive Advanced Solid Tumors
Keywords: claudin18.2; CAR-T; CAR T-cell therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells treatment (Experimental)
  Interventions: Drug: claudin18.2 CAR-T

INTERVENTIONS:
Drug: claudin18.2 CAR-T — injection of CAR T cells

SUMMARY:
The purpose of this clinical trial is to learn if autologous claudin18.2-directed chimeric antigen receptor T-cell (CAR-T) therapy works to treat claudin18.2 positive solid tumors in adults. It will also learn about the safety and efficacy of the autologous claudin18.2 CAR-T cell product.

The main questions it aims to answer are:

1. What CAR-T-related adverse events (AEs) occur within 3 months after the autologous CAR-T cell infusion?
2. What is the Objective Response Rate (ORR), Progression-free survival (PFS), duration of response (DOR), and overall survival (OS)?

Participants will:

1. Undergo leukapheresis for collection of autologous T cells for CAR-T cell manufacturing.
2. May receive lymphodepletion chemotherapy (fludarabine plus cyclophosphamide) for 3 consecutive days if clinically needed.
3. If lymphodepletion chemotherapy is administered, rest for 2 days on Day -2 and Day -1.
4. Receive autologous CAR-T cells infusion on Day 0.
5. Be hospitalized for at least 7 days post-infusion for close safety monitoring and remain within 2 hours of the treatment facility for at least 28 days.
6. Visit the clinic at Day 14, Day 28, then monthly for up to 12 months after CAR-T cells infusion, with continued long-term follow-up for safety and persistence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years at the time of signing the the informed consent form (ICF).
* Pathologically confirmed advanced solid tumor and patients have failed at least 2 prior lines of systemic therapy; or patients with advanced pancreatic cancer who have failed at least 1 prior line of systemic therapy.
* Tumor tissue testing meets the requirement: Positive for Claudin 18.2 (CLDN18.2) by immunohistochemistry (IHC) staining.
* Estimated life expectancy ≥ 12 weeks from the time of screening.
* Presence of measurable tumor lesions in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2 at screening, within 24 hours prior to apheresis, and at baseline.
* Has adequate venous access to allow successful collection of peripheral blood mononuclear cells (PBMCs).
* Meets the specified laboratory test criteria at screening and pre-treatment (see Appendix for detailed parameters). For abnormal laboratory results that do not meet the criteria, a retest is permitted within 1 week; if the retest still fails to meet the criteria, the patient is deemed ineligible for screening.
* Female patients of childbearing potential must have a negative serum pregnancy test at screening and pre-treatment. They must agree to use a highly effective and reliable contraceptive method for 1 year after the last study treatment.
* Male patients who are sexually active with women of childbearing potential must agree to use barrier contraception (unless they have undergone vasectomy) during the study and for 1 year after the last study treatment.
* Voluntarily agrees to participate in the clinical trial, has been fully informed of the study details, signs the ICF, and is willing to comply with and capable of completing all study procedures.

Exclusion Criteria:

* Pregnant or lactating women.
* Serologically positive for human immunodeficiency virus (HIV), Treponema pallidum, or hepatitis C virus (HCV); or positive for Epstein-Barr virus (EBV)-DNA, cytomegalovirus (CMV)-DNA, or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) nucleic acid.
* Presence of any uncontrolled active infection, including but not limited to active tuberculosis and active hepatitis B virus (HBV) infection (defined as HBsAg positive with detectable HBV-DNA).
* Persistent toxicities from prior anti-tumor therapy that have not resolved to Common Terminology Criteria for Adverse Events (CTCAE) grade ≤ 1, except for tolerable events such as alopecia as determined by the investigator.
* Known history of active autoimmune diseases (including but not limited to psoriasis, rheumatoid arthritis) or other conditions requiring long-term immunosuppressive therapy.
* History of hypersensitivity to immunotherapeutic agents or related drugs, history of severe allergies, or hypersensitivity to any component of CAR-T injection.
* Presence of brain metastases or symptoms related to brain metastases.
* Patients at high risk of bleeding or perforation (e.g., active gastrointestinal ulcer, recent gastrointestinal bleeding within 3 months).
* Patients requiring anticoagulant therapy.
* Patients requiring continuous antiplatelet therapy.
* History of organ transplantation or awaiting organ transplantation.
* History of major surgery or significant trauma within 4 weeks prior to apheresis, or planned major surgery during the study period.
* Presence of other serious pre-existing medical conditions that may limit the patient's participation in the study (e.g., severe cardiac, hepatic, or renal dysfunction).
* Assessed by the investigator as unable or unwilling to comply with the study protocol requirements.
* Presence of clinically significant central nervous system (CNS) disease signs or abnormally significant neurological test results.
* Current diagnosis or history of other incurable malignant tumors within the past 3 years, except for in situ cervical cancer or basal cell carcinoma of the skin (which are considered cured after appropriate treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence rate of CAR-T-related adverse events | up to 3 months after CAR-T injection

SECONDARY OUTCOMES:
objective response rate (ORR) | up to 18 months
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Progression-free survival (PFS) | up to 18 months
Duration of response (DOR) | up to 18 months
Overall Survival (OS) | up to 18 months

OTHER OUTCOMES:
AUC of CAR-T cells | up to 2 months after CAR-T injection
  AUCS is defined as the area under the curve in 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided